CLINICAL TRIAL: NCT06142006
Title: A Pilot Study to Test the Feasibility and Acceptability of a Novel Diabetes Staging System in Patient Aligned Care Teams in the Durham VA System
Brief Title: The Diabetes Staging System in Patient Aligned Care Teams
Status: Recruiting | Type: Observational
Sponsor: Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 1746160
Record Dates: First submitted 2023-09-21; First posted 2023-11-21 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Diabetes Staging System (DSS) use among Primary Care Teams — Evaluate the feasibility of using the DSS in PACT clinics to increase SGLT2i and/or GLP-1 agonist use in Veteran DM2 patients with cardiovascular disease

SUMMARY:
The purpose of this study is to examine the feasibility/acceptability of the Diabetes Staging System (DSS) in Patient Aligned Care Teams (PACT) teams and its ability to increase sodium-glucose cotransporter-2 inhibitor (SGLT2i) and glucagon-like-1 peptide (GLP-1) use in Veteran patients with type 2 diabetes and cardiovascular disease and/or chronic kidney disease.

DETAILED DESCRIPTION:
The Diabetes Staging System (DSS) is a novel type 2 diabetes (DM2) staging system patterned after Tumor Node Metastasis (TNM) cancer staging that uses the number of macrovascular and microvascular complications and most recent A1C and glomerular filtration rate (GFR) to determine DSS stage which reflects disease severity. The DSS stage is then linked to specific evidence-based clinical interventions that decrease morbidity and mortality. One of the most important clinical interventions of the DSS is recommending a SGLT2i/GLP-1 agonist in DM2 patients with CVD which helps address the inequity of low overall SGLT2i/GLP-1 use. The DSS has been adapted into a CPRS-DSS template available to all PACT providers within the Durham VA system which could address the racial differences in SGLT2i/GLP-1 agonist use. DSS offers a systematic approach to DM2 care (Stage DM2 -determine medical therapy based on DM2 stage) that has the potential to address inequities related to SGLT2i/GLP-1 overall use and racial differences in use. Primary Care Aligned Teams (PACT) are best positioned to use the DSS because they treat the vast majority of Veteran DM2 patients. This pilot proposal will seek to address inequities in SGLT2i/GLP-1 agonist use within in the VA by examining the feasibility and acceptability of the DSS among 12 different PACT teams within the Durham VA Medical System by measuring its ability to increase SGLT2i/GLP-1 agonist after 6 months of DSS implementation.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* prior history of cardiovascular disease (myocardial infraction, cardiac stents, coronary artery pass, diastolic/systolic heart failure, stroke, carotid endarterectomy, femoral popliteal bypass, abdominal aortic aneurysm)
* prior history of chronic kidney disease (GFR <60, microalbumin creatinine/ratio >30 mg/g - creatinine on 3 separate occasions)
* age 25-75 years
* BMI >27
* diagnosis of type 2 diabetes
* hemoglobin A1C >7.0%
* agreeable to regular visits per study protocol
* access to telephone and reliable transportation and has an assigned PACT provider using a Freestyle Libre 2 or Freestyle lite glucometer to monitor blood sugars or willing to monitor blood sugars during study

Exclusion Criteria:

* age >75,
* A1C <7%
* GFR <30
* pregnant
* breast feeding
* prior history of pancreatitis will lead to avoidance of GLP-1 agonist therapy but not SGLT2i
* prior history of gastroparesis, dysphagia will lead to avoidance of GLP-1 agonist therapy but not SGLT2i
* history of thyroid cancer/multiple endocrine neoplasia/thyroid nodules/medullary thyroid cancer (contraindication to Liraglutide) will lead to avoidance of GLP-1 agonist therapy but not SGLT2i
* history of gallstones will lead to avoidance of GLP-1 agonist therapy but not SGLT2i history of hyperoxaluria or calcium oxalate nephrolithiasis will lead to avoidance of GLP-1 agonist therapy but not SGLT2i
* history of Roux-en-Y gastric bypass or gastric sleeve or any other bariatric procedure will lead to avoidance of GLP-1 agonist therapy but not SGLT2i
* type 1 diabetes
* any gastrointestinal condition causing malabsorption (including but not limited to inflammatory bowel disease, celiac sprue) will lead to avoidance of GLP-1 agonist therapy but not SGLT2i
* prior history of urinary tract infections will lead to avoidance of SGLT2i but not GLP-1 agonist therapy
* prior h/o recurrent yeast infections will lead to avoidance of SGLT2i but not GLP-1 agonist therapy
* uncircumcised male will lead to avoidance of SGLT2i but not GLP-1 agonist therapy prior h/o toe or lower extremity amputations will lead to avoidance of SGLT2i but not GLP-1 agonist therapy
* active diabetic foot ulcers or osteomyelitis will lead to avoidance of SGLT2i but not GLP-1 agonist therapy
* unwilling or unable to complete scheduled testing
* any serious and/or unstable medical, psychiatric, or other condition(s) that prevents the patient from providing informed consent or complying with the study
* organ transplantation or those on immunosuppressants
* chronic anticoagulation
* recent myocardial infarction, unstable angina, stroke, coronary artery bypass or transient ischemia attacks in the past 6 months
* chronic prednisone use
* deep vein thrombosis in past 6 months
* active malignancy-unstable psychiatric condition including active or current suicidal ideation
* Enrolled in another research study related to diet and/or physical activity

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible subjects within each PACT team will be identified retrospectively at baseline to by the study coordinator using inclusion/exclusion criteria noted below. There is no specific number of subjects that will be enrolled rather we will make a determination of % of Veterans with DM2 and CVD who are on SGLT2i/GLP-1 agonist at baseline and after 6 months of DSS use by the participating PACT teams. Veteran patients will not require consent because SGLT2i/GLP-1 agonist is standard of care in DM2 with CV disease patients.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
SGLT2i and/or GLP-1 agonist use after DSS EHR template use | Baseline and 6 months after DSS implementation
  Percentage of Caucasian and African American DM2 Veteran patients with CVD who are on SGLT2i and/or GLP-1 agonist at baseline and 6 months after provider DSS EHR template use.

SECONDARY OUTCOMES:
Weight | Baseline and 6 months after DSS implementation
  Measured in pounds
Blood pressure | Baseline and 6 months after DSS implementation
  Measures systolic and diastolic blood pressure in mmHG
Hemoglobin A1C | Baseline and 6 months after DSS implementation
  Measures average blood sugars control over the past 3 months
GFR | Baseline and 6 months after DSS implementation
  Measures glomerular filtration rate

CONTACTS AND LOCATIONS:
Overall Officials: Moahad S Dar, MD, Principal Investigator — Department of Veterans Affair, Durham VAHCS
Locations (1):
- Greenville VA Health Care Center, 401 Moye Blvd, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dar MS, Beg SA. TNM cancer staging: can it help develop a novel staging system for type 2 diabetes? Diabetes Metab Syndr Obes. 2018 Nov 28;11:845-853. doi: 10.2147/DMSO.S179963. eCollection 2018. PMID 30568472
- [Background] Dar MS, Wanner C, Marx N, Ofstad AP, Mattheus M, Kaspers S, Beg SA. Cardiovascular outcomes trial data from EMPA-REG OUTCOME, CAROLINA and CARMELINA: Assessment of a novel staging system for type 2 diabetes. Diabetes Obes Metab. 2023 May;25(5):1372-1384. doi: 10.1111/dom.14989. Epub 2023 Mar 6. PMID 36700391